CLINICAL TRIAL: NCT06454890
Title: An Investigator-initiated Trial Evaluating the Efficacy and Safety of Anti-Trop2 Universal CAR-NK(U-CAR-NK) Cells Therapy Combined With Chemotherapy for Relapsed/Refractory Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Clinical Study of Trop2 CAR-NK in the Treatment of Relapsed/Refractory Non-Small Cell Lung Cancer (NSCLC)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Qiming Wang, Professor, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHH-101-NSCLC
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Non-Small Cell Lung Cancer NSCLC
Keywords: CAR-NK, TROP2, NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-Trop2 CAR-NK cell therapy group (Experimental): chemotherapy followed by Trop2 CAR-NK infusion
  Interventions: Biological: Anti-Trop2 CAR-NK cell

INTERVENTIONS:
Biological: Anti-Trop2 CAR-NK cell — chemotherapy followed by Trop2 CAR-NK infusion

SUMMARY:
It is a single-center, open-labeled, single-arm, non-randomized investigator-initiated trial evaluating the efficacy and safety of anti-Trop2 U-CAR-NK Cells Therapy combined with Chemotherapy for Relapsed/Refractory Non-Small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
Who can participate? Patients who were diagnosed with Non-Small Cell Lung Cancer and tumor cells expressing Trop2.

How to conduct this study? This study is an interventional clinical study. The intervention in the trial is anti-Trop2 U-CAR-NK cells. The administration time is 5 days after chemotherapy. Patients were then evaluated efficacy and safety until 3 years after U-CAR-NK cells infusion.

What are the possible benefits and risks of participating? Benefits: The effect of anti-tumor of NK cells may be used to disease control.

Risks: Subjects may have adverse reactions to the treatment. These adverse reactions may include abnormal liver injury, fever, and possibly other unknown adverse reactions.

Where is the study run? Henan Cancer Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-79, male and female;
2. Predicted survival ≥12 weeks;
3. ECOG score 0-1;
4. Diagnosed with Stage IIIB-IV non-small cell lung cancer (NSCLC) through imaging, histological, and/or cytological examinations
5. For patients with negative driver genes (EGFR/ALK/ROS-1/BRAF V600E/MET exon 14 mutation/NTRK), failed first-line PD-1/PD-L1 immunotherapy combined with platinum-based doublet chemotherapy; For patients with EGFR-sensitive mutations (19del, 21L858R, 18exonG719X, 20exonS768I, 21exonL861Q), they must meet one of the following requirements: a) Failed treatment with 1st or 2nd generation EGFR-TKI, and histologically confirmed T790M mutation negative after treatment failure; b) Failed treatment with 3rd generation EGFR-TKI regardless of T790M mutation status; For patients with other driver genes positive besides EGFR mutation and have approved first-line targeted therapies, failed first-line targeted therapy;
6. Have at least one measurable tumor lesion according to RECIST 1.1;
7. The tumor tissue sample (previous or fresh) shows at least 50% weak positive expression of Trop2 protein;
8. Have adequate organ and bone marrow function, defined as follows:

   Blood routine: Absolute neutrophil count (ANC) ≥ 1.5×109/L, platelet (PLT) ≥ 100×109/L, hemoglobin (Hb) ≥ 90g/L; Liver function: Bilirubin < 1.5 times the upper limit of normal (ULN), alkaline phosphatase (ALP), aspartate aminotransferase (AST), and alanine aminotransferase (ALT) < 2.5 times ULN (in case of liver metastasis, ALP, AST, and ALT < 5 times ULN are allowed); Renal function: Creatinine clearance rate (CCR) ≥ 60 mL/min (using the standard Cockcroft-Gault formula);
9. For women: surgically sterilized, postmenopausal patients, or those who agree to use a medically accepted contraceptive method (such as intrauterine device, contraceptive pills, or condoms) during and for 6 months after the study treatment period; serum or urine pregnancy test must be negative within 7 days before study enrollment, and must be non-lactating; For men: surgically sterilized or those who agree to use a medically accepted contraceptive method during and for 6 months after the study treatment period.

Exclusion Criteria:

1. Severe infection;
2. Clinically active brain or meningeal metastasis, defined as untreated and symptomatic, or requiring steroids or anticonvulsant therapy to control related symptoms. For asymptomatic brain metastasis subjects, if they have been stable for at least 4 weeks in imaging and neurologically after receiving targeted therapy for brain metastasis, and are on a stable or reduced dose of steroids equivalent to ≤10 mg/day of prednisone, they may be included in the study;
3. Organic heart disease, cardiac insufficiency, heart block above grade II, myocardial infarction within 6 months;
4. Active autoimmune disease;
5. Interstitial lung disease;
6. Active hepatitis B (Hepatitis B surface antigen (HBsAg) positive, HBV-DNA testing required; HBV-DNA ≥500 IU/mL or higher than the lower limit of detection, whichever is higher) or hepatitis C (Hepatitis C antibody positive and HCV-RNA higher than the lower limit of detection);
7. Positive human immunodeficiency virus (HIV) test or history of acquired immunodeficiency syndrome (AIDS); known active syphilis infection;
8. Pregnancy or lactation;
9. Patients with a tendency to bleed, including acute gastrointestinal bleeding, nasal bleeding, hemoptysis, as well as persistent bleeding disorders or coagulation disorders;
10. Patients who have used anti-tumor drugs other than immunotherapy within 3 weeks;

12. Multiple primary malignancies within 3 years prior to enrollment, except for fully resected non-melanoma skin cancer (e.g., resected basal or squamous cell skin cancer), radically treated carcinoma in situ (e.g., cervical or breast carcinoma in situ), other radically treated solid tumors (e.g., superficial bladder cancer), or contralateral breast cancer; 13. History of allergy to any component of the study drug; 14. Other situations that the investigator deems unsuitable for participation in the study, or other situations that may affect the analysis of the clinical study results.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety by Common Terminology Criteria for Adverse Events (CTCAE) V5.0 | Up to 1 year
  The type, frequency, severity, and duration of adverse events as a result of Trop2 CAR-NK cells infusion will be summarized.
Objective Response Rate (ORR) | up to 1 year.
  Per Response Evaluation Criteria in Solid Tumours (RECIST 1.1) assessed by MRI or CT. ORR defined as the proportion of patients in whom a complete response (CR) or partial response (PR) is observed as best overall response, prior to progression or further anti-cancer therapy.

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to 1 year.
  Disease control rate (DCR) defined as the proportion of patients in whom a CR or PR or stable disease (SD) (per RECIST 1.1, SD assessed at least 6 weeks after the first dose) is observed as best overall response.
Overall survival (OS) | up to 3 years.
  To determine the anti-tumor effectivity

CONTACTS AND LOCATIONS:
Overall Officials: Qiming Wang PhD, Principal Investigator — Henan Cancer Hospital

IPD SHARING:
Plan to Share IPD: No